CLINICAL TRIAL: NCT03914976
Title: Association of the Arteriovenous Difference in Carbon Dioxide and Its Relation to the Difference in Arteriovenous Oxygen Content With the Occurrence of Postoperative Complication
Acronym: CARBODAV
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0041; 2019-A00323-54 (Other: ANSM)
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Surgery--Complications
Keywords: high-risk digestive surgery; intensive care unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — It was estimated that there is between 40 and 60 ml of blood taken during this kind of intervention and in 24-hour postoperative intervention .
  The completion of the study should result in an increase in blood volume taken from 5 to 10 mL
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient who will have a high risk digestive surgery: patient who will have a high risk digestive surgery: esophagectomy, major hepatectomy> 3 segments, duodeno cephalic pancreatectomy
  Interventions: Procedure: patient having to undergo a high risk programmed digestive surgery

INTERVENTIONS:
Procedure: patient having to undergo a high risk programmed digestive surgery — The objective is to determine if there is an association between the mean intraoperative values and within 24 hours postoperative ΔPCO2 and the occurrence of major post-operative complications at day 28 in high-risk surgery (major hepatectomy, esophagectomy or duodeno- cephalic pancreatectomy)

SUMMARY:
Intra-operative hemodynamic management in high-risk surgery is a priority for the anesthesiologist. The current strategy is based on the continuous measurement of cardiac output and its maximization by vascular filling has many limitations: invasiveness, measurement difficulties, impaired performance, imperative surgical restriction of filling, lack of evaluation of flow rate and metabolic needs. Biomarkers may be able to detect early an inadequacy between cardiac output and tissue oxygen requirements, venous saturation with oxygen (ScvO2) and arteriovenous difference in partial pressure of carbon dioxide (ΔPCO2) as well as the appearance of cellular hypoxia (lactate and arteriovenous difference in partial pressure of carbon dioxide/arteriovenous difference in oxygen) (ΔPCO2) / DAVO2). Moreover, the medical literature remains poor on the evaluation of these markers in per-operative context all the more for ΔPCO2 and ΔPCO2 / DAVO2. It seems interesting to evaluate the potential of these tools, in patients with major surgery and at high risk (major hepatectomy, oesophagectomy and duodeno-pancreatectomy), to predict the risk of postoperative complications, especially since surgery involves a restrictive vascular filling strategy that may be potentially deleterious to the patient.

ELIGIBILITY:
Inclusion Criteria:

Major patient

Patient eligible for a high risk scheduled gastrointestinal surgery from:

* Esophagectomy
* Major hepatectomy (≥ 3 segments)
* Cephalic duodeno-pancreatectomy Patient with an arterial catheter and a central venous line in superior vena cava.

Patient hospitalized post-operatively in intensive care unit as agreed in consultation with preoperative anesthesia.

Exclusion Criteria:

* Pregnant or lactating patients
* Patient with an unstable acute condition at the time of surgery (acute heart, respiratory or renal failure, severe sepsis or septic shock, hemorrhagic shock)
* Patient opposing his participation in the study
* Patient protected by law (guardianship)
* Patient deprived of liberty
* Patient with a contraindication to the establishment of a central venous route in superior vena cava territory or a radial or femoral arterial catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study concerns patients operated for a high-risk digestive surgery, hospitalized postoperatively in intensive care unit (agreed in anesthesia consultation). These patients will also need to have an arterial catheter and a central venous line in the superior vena cava
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
mean intraoperative PCO2 values | during surgery
  PCO2 values will be collected every 2 hours during surgery
mean postoperative PCO2 values | within 24 hours after surgery
post-operative complications | 28 days after surgery
  post-operative complications of grade III or greater according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu GAZON, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Derived] Guilherme E, Delignette MC, Pambet H, Lebreton T, Bonnet A, Pradat P, Boucheny C, Guichon C, Aubrun F, Gazon M. PCO2 gap, its ratio to arteriovenous oxygen content, ScvO2 and lactate in high-risk abdominal surgery patients: An observational study. Anaesth Crit Care Pain Med. 2022 Apr;41(2):101033. doi: 10.1016/j.accpm.2022.101033. Epub 2022 Feb 14. PMID 35176527